CLINICAL TRIAL: NCT02006628
Title: A Double-blind, Randomised, Placebo-controlled, Parallel Group Study of GWP42003 as Adjunctive Therapy in the First Line Treatment of Schizophrenia or Related Psychotic Disorder
Brief Title: A Study of GWP42003 as Adjunctive Therapy in the First Line Treatment of Schizophrenia or Related Psychotic Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWAP1241; 2013-000212-22 (EudraCT Number)
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Schizophrenia; Schizophrenia-related Psychotic Disorder
Keywords: GWP42003; Cannabinoids; Schizophrenia; CBD; Cannabidiol
MeSH Terms: conditions — Schizophrenia | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GWP42003 1000 milligrams (mg)/day (Active Comparator): Participants received GWP42003 (100 mg/milliliter [mL]), 5 mL twice daily (BID) administered orally, 5 mL in the morning and 5 mL in the evening for 6 weeks.
  Interventions: Drug: GWP42003
- Placebo (Placebo Comparator): Participants received placebo (0 mL cannabidiol [CBD]), volume matched to the 5 mL BID dose level, administered orally, 5 mL in the morning and 5 mL in the evening for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo oral solution (0 milligrams [mg]/mL CBD) contained the excipients sesame oil, ethanol, sucralose, and strawberry flavoring.
  Other Names: Placebo control
  Arms: Placebo
Drug: GWP42003 — GWP42003 was an oral solution containing 100 mg/mL CBD dissolved in the excipients sesame oil, ethanol, sucralose and strawberry flavoring.
  Other Names: Cannabidiol
  Arms: GWP42003 1000 milligrams (mg)/day

SUMMARY:
A study to compare the change in symptom severity in participants with schizophrenia or related psychotic disorder when treated with GWP42003 or placebo in conjunction with existing anti-psychotic therapy over a period of six weeks.

DETAILED DESCRIPTION:
This eight-week (six-week treatment period and two-week follow-up), multi-centre, double-blind, randomized, placebo-controlled, parallel group study aimed to determine the efficacy, safety and tolerability of GWP42003 in participants with schizophrenia or a related psychotic disorder.

Eligible participants entered the study at a Screening and Randomization Visit (Day 1), where eligibility was established. Once all inclusion and exclusion criteria were reviewed, participants were randomized to receive either GWP42003 or placebo in conjunction with their prescribed anti-psychotic medications and began treatment on Day 1 as instructed. Assessments were performed on Days 8, 22, and 43. A safety follow-up visit was conducted on Day 57.

ELIGIBILITY:
Inclusion Criteria (all must be fulfilled):

* Participant gave written informed consent for participation in the study and did not require involuntary treatment.
* Participant was male or female aged 18 to 65 years.
* Participant was able (in the investigator's opinion) and willing to comply with all study requirements.
* Participant was diagnosed with schizophrenia or a related psychotic disorder (such as schizoaffective or schizophreniform disorder) as defined by the Diagnostic and Statistical Manual of Mental Disorders Version 4.
* Participant was treated for a minimum of four-weeks and was on a stable dose of his or her current anti-psychotic (AP) medication.
* Participant showed the capacity to respond at least partially to first line AP medication in the opinion of the investigator.
* Participant remained stable on his or her dose of AP and concomitant medications for the duration of the study, in the opinion of the investigator.
* Participant was willing for his or her name to be notified to the responsible authorities for participation in this study, as applicable in individual countries.
* Participant was willing to allow his or her primary care practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria (any of the following):

* Participant had any known or suspected hypersensitivity to cannabinoids or any of the excipients of the Investigational Medicinal Product (IMP).
* Participant had a Positive and Negative Symptom Scale total score of <60 at Day 1.
* Participant presented with a current clinical picture and/or history that is consistent with:

  i. delirium or dementia. ii. acute drug induced psychosis. iii. bipolar disorder.
* Participant was taking more the one AP medication during the study.
* Female participants of child bearing potential and male participants whose partner was of child bearing potential, unless willing to ensure that they or their partner used effective contraception, for example, oral contraception, double barrier, intra-uterine device, during the study and for three months thereafter (a male condom was not used in conjunction with a female condom).
* Female participant who was pregnant, lactating, or planning pregnancy during the course of the study and for three months thereafter.
* Participants who had received an IMP within 30 days prior to the screening visit.
* Participants who had any other significant disease or disorder which, in the opinion of the investigator, either put the participant at risk because of participation in the study, or may have influenced the result of the study, or the participant's ability to participate in the study.
* Participant had any abnormalities following a physical examination that, in the opinion of the investigator, prevented the participant from safe participation in the study.
* Participant was unwilling to abstain from donation of blood during the study.
* Participant had travelled outside the country of residence during the study.
* Participant previously randomized into this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-02-25 (Actual); Primary Completion 2015-01-08 (Actual); Study Completion 2015-01-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Poland (6):
  - Czeladź
  - Gdansk
  - Kielce
  - Lublin
  - Tychy
  - Wroclaw
- Romania (4):
  - Bucharest
  - Sibiu
  - Târgovişte
  - Târgu Mureş
- United Kingdom (3):
  - Chertsey
  - Coventry
  - London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGuire P, Robson P, Cubala WJ, Vasile D, Morrison PD, Barron R, Taylor A, Wright S. Cannabidiol (CBD) as an Adjunctive Therapy in Schizophrenia: A Multicenter Randomized Controlled Trial. Am J Psychiatry. 2018 Mar 1;175(3):225-231. doi: 10.1176/appi.ajp.2017.17030325. Epub 2017 Dec 15. PMID 29241357

RESULTS

PARTICIPANT FLOW:
Groups:
- GWP42003 1000 Milligram (mg)/Day: Participants received GWP42003 (100 mg/milliliter [mL]), 5 mL twice daily (BID) administered orally, 5 mL in the morning and 5 mL in the evening for 6 weeks.
Period: Overall Study
Arm/Group | GWP42003 1000 Milligram (mg)/Day | Placebo
Started | 43 | 45
Received at Least 1 Dose of Study Drug (Safety analysis set) | 43 | 45
Intention to Treat (ITT) Analysis Set (Provided informed consent, randomized, took at least 1 dose of IMP, had post-baseline efficacy data) | 42 | 44
Completed | 40 | 43
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set: Participants who provided informed consent, were randomized to 1 of the treatment groups, and took at least 1 dose of investigational medicinal product (IMP).
Groups:
- GWP42003 1000 mg/Day: Participants received GWP42003 (100 mg/mL), 5 mL BID administered orally, 5 mL in the morning and 5 mL in the evening for 6 weeks.
- Placebo: Participants received placebo (0 mL CBD), volume matched to the 5 mL BID dose level, administered orally, 5 mL in the morning and 5 mL in the evening for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | GWP42003 1000 mg/Day | Placebo | Total
Number analyzed (Participants) | 43 | 45 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (12.49) | 40.8 (11.00) | 40.8 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 22 | 37
  Male | 28 | 23 | 51

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline To End Of Treatment (Day 43) In Positive And Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS was a 30-item medical scale completed by a trained rater that assessed the positive and negative symptoms of schizophrenia as well as symptoms of general psychopathology. The PANSS Total score was derived from the sum of the 30 items, which were rated on a 7-point scale, where 1 = absent and 7 = extreme. The total score is the summed total for each of the PANSS positive symptom ('P'), negative symptom ('N'), general psychopathology symptom ('G') scores and could range from 30 to 210 points, with lower scores equating to milder severity of symptoms, that is, closer to psychologically normal.
Time Frame: Day 1 through Day 43
Population: ITT analysis set: all participants who provided informed consent, were randomized to 1 of the treatment groups, took at least 1 dose of IMP, and had post-baseline efficacy data. One placebo participant with a PANSS Total score <60 at Day 1 and 1 GWP42003 participant with no post-baseline efficacy data were excluded from the ITT analysis set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GWP42003 1000 mg/Day | Placebo
Number analyzed (Participants) | 42 | 44
score on a scale
  Baseline score | 79.3 (12.45) | 80.6 (14.90)
  End of Treatment score | 68.1 (14.79) | 71.9 (15.49)
  Change from baseline | -11.2 (7.87) | -8.8 (8.87)
Statistical Analysis 1: Comparison: GWP42003 1000 mg/Day vs Placebo; Test type: Superiority; p = 0.1332, ANCOVA; Change from baseline as the response variable, treatment as fixed effect, and individual baseline subscore and age as covariates; Treatment difference (GWP42003-placebo) = -2.8, 95% CI 2-sided [-6.5 to 0.9]

2. Primary Outcome: Percentage Of PANSS Total Score Responders At End Of Treatment (Day 43)
Description: The percentage of PANSS treatment responders, defined as participants with ≥20% improvement in PANSS Total score between baseline and End of Treatment, is presented. The percentage of participants was calculated by dividing the number of participants with a ≥20% improvement in PANSS Total score (yes) by the total number of participants.
Time Frame: Day 1 through Day 43
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003 1000 mg/Day | Placebo
Number analyzed (Participants) | 42 | 44
Participants
  Yes | 12 | 6
  No | 30 | 38
Statistical Analysis 1: Comparison: GWP42003 1000 mg/Day vs Placebo; Test type: Superiority; p = 0.0896, Regression, Logistic; Responder (yes/no) is the dependent variable with treatment included as factor and age and baseline P, G, and N scores included as covariates; Odds Ratio (OR) = 2.62, 95% CI 2-sided [0.86 to 8.00]

3. Primary Outcome: Change From Baseline To The End Of Treatment (Day 43) In PANSS 'P' Score
Description: The PANSS 'P' scale measured the severity of positive symptoms, including delusions, conceptual disorganization, hallucinations, hyperactivity, grandiosity, suspiciousness/persecution, and hostility. Individual items were rated on a 7-point scale, where 1 = absent and 7 = extreme. The total 'P' score could range from 7 to 49 points, with lower scores equating to milder severity of symptoms, that is, closer to psychologically normal.
Time Frame: Day 1 through Day 43
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GWP42003 1000 mg/Day | Placebo
Number analyzed (Participants) | 42 | 44
score on a scale
  Baseline score | 18.0 (3.89) | 17.5 (3.29)
  End of Treatment score | 14.8 (4.01) | 15.7 (3.73)
  Change from Baseline | -3.2 (2.60) | -1.7 (2.76)
Statistical Analysis 1: Comparison: GWP42003 1000 mg/Day vs Placebo; Test type: Superiority; p = 0.0188, ANCOVA; Treatment difference (GWP42003-placebo) = -1.4, 95% CI 2-sided [-2.5 to -0.2]

4. Primary Outcome: Change From Baseline To The End Of Treatment (Day 43) In PANSS 'N' Score
Description: The PANSS 'N' scale measured the severity of negative symptoms, including blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, and stereotyped thinking. Individual items were rated on a 7-point scale, where 1 = absent and 7 = extreme. The total 'N' score could range from 7 to 49 points, with lower scores equating to milder severity of symptoms, that is, closer to psychologically normal.
Time Frame: Day 1 through Day 43
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GWP42003 1000 mg/Day | Placebo
Number analyzed (Participants) | 42 | 44
score on a scale
  Baseline score | 22.6 (5.04) | 23.4 (5.11)
  End of Treatment score | 19.9 (5.32) | 20.5 (5.22)
  Change from Baseline | -2.7 (3.55) | -2.9 (3.06)
Statistical Analysis 1: Comparison: GWP42003 1000 mg/Day vs Placebo; Test type: Superiority; p = 0.9647, ANCOVA; Treatment difference (GWP42003-placebo) = 0.0, 95% CI 2-sided [-1.3 to 1.4]

5. Primary Outcome: Change From Baseline To The End Of Treatment (Day 43) In PANSS 'G' Score
Description: The PANSS 'G' scale measured the severity of general psychopathology symptoms, including somatic concern, anxiety, guilt feelings, tension, mannerisms and posturing, depression, motor retardation, uncooperativeness, unusual thought content, disorientation, poor attention, lack of judgement and insight, disturbance of violation, poor impulse control, preoccupation, and active social avoidance. Individual items were rated on a 7-point scale, where 1 = absent and 7 = extreme. The total 'G' score could range from 16 to 112 points, with lower scores equating to milder severity of symptoms, that is, closer to psychologically normal.
Time Frame: Day 1 through Day 43
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GWP42003 1000 mg/Day | Placebo
Number analyzed (Participants) | 42 | 44
score on a scale
  Baseline score | 38.7 (6.71) | 39.7 (8.95)
  End of Treatment score | 33.4 (7.69) | 35.6 (9.04)
  Change from Baseline | -5.3 (4.34) | -4.1 (4.78)
Statistical Analysis 1: Comparison: GWP42003 1000 mg/Day vs Placebo; Test type: Superiority; p = 0.1963, ANCOVA; Treatment difference (GWP42003-placebo) = -1.3, 95% CI 2-sided [-3.2 to 0.7]

6. Primary Outcome: Change From Baseline To The End Of Treatment (Day 43) In The Scale For The Assessment Of Negative Symptoms (SANS)
Description: The SANS assessed 5 symptom complexes to obtain clinical ratings of negative symptoms in participants with schizophrenia or related psychotic disorder. Symptom complexes were affective blunting, alogia (impoverished thinking), avolition/apathy, anhedonia/asociality, and disturbance of attention. Assessments were conducted on a 6-point scale (0 = not at all; 5 = severe). The total score could range from 0 to 125 points, with lower scores equating to milder severity of symptoms, that is, closer to psychologically normal.
Time Frame: Day 1 through Day 43
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GWP42003 1000 mg/Day | Placebo
Number analyzed (Participants) | 42 | 44
score on a scale
  Baseline score: number analyzed (Participants) | 42 | 43
  Baseline score | 52.8 (17.10) | 55.3 (16.24)
  End of Treatment score | 43.6 (16.54) | 48.4 (15.75)
  Change from Baseline | -9.1 (13.09) | -6.3 (8.54)
Statistical Analysis 1: Comparison: GWP42003 1000 mg/Day vs Placebo; Test type: Superiority; p = 0.1167, ANCOVA; Treatment difference (GWP42003-placebo) = -3.5, 95% CI 2-sided [-7.9 to 0.9]

7. Primary Outcome: Change From Baseline To The End Of Treatment (Day 43) In The Clinical Global Impression Severity Scale (CGI-S)
Description: The CGI-S was a 7-point scale that required the clinician to rate the severity of a participant's illness at the time of assessment, relative to the clinician's past experience of participants who had the same diagnosis. Considering total clinical experience, participants were assessed on severity of mental illness at the time of rating on the following scale: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; or 7 = extremely ill. Lower scores equated to milder severity of symptoms, that is, closer to psychologically normal.
Time Frame: Day 1 through Day 43
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GWP42003 1000 mg/Day | Placebo
Number analyzed (Participants) | 42 | 44
score on a scale
  Baseline score | 4.0 (0.70) | 4.0 (0.65)
  End of Treatment score | 3.5 (1.09) | 3.8 (0.78)
  Change from Baseline | -0.5 (0.74) | -0.3 (0.49)
Statistical Analysis 1: Comparison: GWP42003 1000 mg/Day vs Placebo; Test type: Superiority; p = 0.0443, ANCOVA; Treatment difference (GWP42003-placebo) = -0.3, 95% CI 2-sided [-0.5 to 0.0]

8. Primary Outcome: Clinical Global Impression Improvement Scale (CGI-I) Values At Day 8 And End Of Treatment (Day 43)
Description: The CGI-I was a 7-point scale that required the clinician to assess how much a participant's illness had improved or worsened relative the first assessment at the beginning of the intervention. This was rated on the following scale: 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; or 7 = very much worse. Lower scores equated to improvement of symptoms.
Time Frame: Day 8 through Day 43
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GWP42003 1000 mg/Day | Placebo
Number analyzed (Participants) | 42 | 44
score on a scale
  Day 8 score: number analyzed (Participants) | 40 | 43
  Day 8 score | 3.6 (0.50) | 3.8 (0.56)
  End of Treatment score | 2.9 (0.89) | 3.4 (0.87)
Statistical Analysis 1: Comparison: GWP42003 1000 mg/Day vs Placebo; Test type: Superiority; p = 0.0182, ANCOVA; Treatment difference (GWP42003-placebo) = -0.5, 95% CI 2-sided [-0.8 to -0.1]

9. Primary Outcome: Change From Baseline To The End Of Treatment (Day 43) In Brief Assessment Of Cognition In Schizophrenia (BACS) Score
Description: The BACS was an instrument used to assess the aspects of cognition found to be most impaired and most strongly correlated with outcome in participants with schizophrenia or related psychotic disorder. The BACS consisted of 6 domains: verbal memory (score range 0 to 75), working memory (score range 0 to 28), motor speed (score range 0 to 100), verbal fluency (score > 0, with no set maximum value), attention and speed of information processing (score range 0 to 110), and executive functions (score range 0 to 22). A score was obtained for each of the 6 domains. A composite summary score was then calculated as the arithmetic mean of the unweighted scores from the 6 domains. While there was not an upper limit on the composite score, overall, an increase in score was indicative of an improvement in cognition.
Time Frame: Day 1 through Day 43
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GWP42003 1000 mg/Day | Placebo
Number analyzed (Participants) | 42 | 44
score on a scale
  Baseline score | 32.21 (6.042) | 32.91 (7.158)
  End of Treatment score: number analyzed (Participants) | 41 | 44
  End of Treatment score | 35.73 (6.981) | 35.05 (7.310)
  Change from Baseline: number analyzed (Participants) | 41 | 44
  Change from Baseline | 3.48 (3.031) | 2.14 (3.442)
Statistical Analysis 1: Comparison: GWP42003 1000 mg/Day vs Placebo; Test type: Superiority; p = 0.0677, ANCOVA; Treatment difference (GWP42003-placebo) = 1.31, 95% CI 2-sided [-0.10 to 2.72]

ADVERSE EVENTS:
Time Frame: Day 1 through Day 57
Description: Safety analysis set: all participants who provided informed consent, were randomized to treatment, and took at least 1 dose of IMP.
Arm/Group | GWP42003 1000 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 0/43 | 1/45
Other Adverse Events (participants affected / at risk) | 8/43 | 10/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003 1000 mg/Day (N=43) | Placebo (N=45)
Schizophrenia (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003 1000 mg/Day (N=43) | Placebo (N=45)
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 3 | 0
Headache (Nervous system disorders) | 3 | 4
Somnolence (Nervous system disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days